CLINICAL TRIAL: NCT01207778
Title: Brain Imaging and Developmental Follow up of Infants Treated With Erythropoietin
Acronym: BRITE
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-153; R01HD059856 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2022-05

CONDITIONS: Prematurity
Keywords: brain; development; erythropoietin; neuroprotection; MRI
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- preterm ESA recipients: Former preterm infants 500-1250 grams who received erythropoietin (400 units/kg 3x/week) or darbepoetin (10 micrograms/kg 1x/week), from the first week of life through 35 weeks corrected gestation
- preterm controls: Former preterm infants 500-1250 grams who received placebo (sham dosing), from first week of life through 35 weeks corrected gestation
- term controls: Former term infants with normal delivery

SUMMARY:
Approximately 60,000 premature infants are born each year who weigh less than 1,500 grams,many of whom sustain brain damage because of their prematurity. This study is designed to evaluate the long-term developmental effects of one promising neuroprotective treatment,erythropoietin (Epo), when given in the neonatal period. Using detailed neurodevelopmental testing and state-of-the-art brain imaging, we hope to determine whether this is an effective treatment to prevent brain injury associated with prematurity, and to lay the groundwork for further studies to improve the developmental outcome of infants delivered prematurely.

DETAILED DESCRIPTION:
Over twelve percent of infants born less than 1,500 grams (VLBW) sustain brain injury with subsequent developmental delay. Although various neuroprotective strategies have been evaluated, none have been successful. One promising intervention is the use of recombinant erythropoietin (Epo, also known as an erythropoiesis stimulating agent, or ESA). In addition to stimulating red cell production, Epo has been shown to be protective in the developing brain in animal models. We have preliminary data suggesting its efficacy when used in VLBW infants, who are at risk of requiring transfusions, and who are also at risk for brain hemorrhage, hypoxicischemic brain injury, and developmental delay. We are currently performing a multicentered study evaluating hematopoietic and short term developmental effects of ESAs in preterm infants randomized to receive Epo, Darbepoetin alfa (a longer acting ESA), or placebo/ control for the first 10 weeks of age (NCT00334737). The first enrolled infants will reach 42-48 months in January, 2010. While that study evaluates the safety and general short-term developmental effects of ESAs, there is an unprecedented opportunity to study long term effects of ESA in significant detail, including evaluating the long term developmental effects and the underlying mechanism of neurologic improvement with state of the art neuroimaging. This proposal seeks to evaluate longitudinal, long-term developmental effects and underlying neurologic mechanisms of ESAs administered to VLBW infants in the first 10 weeks of life. Our specific hypotheses are:

1) ESAs administered to preterm infants during the neonatal period improve long-term neurodevelopmental outcome, 2) ESAs affect regional brain structure, neurochemistry and neurologic organization as reflected in magnetic resonance (MR) imaging, and 3) the blood level of ESA correlates with MR imaging and neurodevelopmental outcome. To test these hypotheses, neurodevelopmental outcome will be assessed through a comprehensive neurodevelopmental assessment at two time points: 42-48 months, and 66-72 months (WPSSI III, Early Child Assessment, Executive Categorization Battery). Brain imaging will be performed concurrent with developmental assessments and includes measures of volume (high resolution volumetric analysis), neurochemistry (magnetic resonance spectroscopy) and regional cerebral blood flow (arterial spin labeling). This study is highly clinically relevant due to the long-term developmental and imaging follow up studies that are part of the design, significantly increasing our ability to determine if developmental, functional and anatomical differences exist in infants randomized to ESAs, a relatively new interventional strategy used in preterm infants. This proposal addresses our long-term goal of developing effective treatment strategies for disorders associated with prematurity through an improved understanding of brain-behavioral relationships.

ELIGIBILITY:
Inclusion Criteria (preterm):

* birth weight 500-1,250 grams, gestational age ≤32 weeks
* hematocrit ≤55%
* ≤48 hours of age
* expected to survive greater than 72 hours
* consent signed by parent or guardian

Inclusion Criteria (term):

Former term born infants will be eligible if they have not experienced any episodes of hypoxia, hypoglycemia, hyperbilirubinemia, prenatal drug exposure, or sepsis.

Exclusion Criteria (former preterms):

* hemorrhagic or hemolytic disease
* major congenital anomalies (such as trisomy 13, 18 or 21)
* major neurologic abnormality such as hydrocephalus or meningomyelocele
* complex congenital heart disease
* receiving Epo or are enrolled in an Epo study
* evidence of disseminated intravascular coagulation
* clinical seizures are present
* congenital thrombotic disease is suspected
* systolic blood pressures >100 mm Hg (while not on pressor support) Infants with minor anomalies such as clinodactyly, single umbilical vessel or patent ductus are not excluded

Exclusion criteria (term):

hypoxia, hypoglycemia, hyperbilirubinemia, prenatal drug exposure, or sepsis

Ages: 36 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants previously enrolled in NCT00334737, a randomized masked study of darbepoetin administration in preterm infants, are eligible for the study. In addition we will enroll term infants matched for age, gender and ethnicity to the preterm group to serve as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2010-03; Primary Completion 2016-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin K Ohls, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - MIND Research Network, Albuquerque, New Mexico
  - UNM, Albuquerque, New Mexico
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Plan to submit data if possible for meta analyses

REFERENCES:
- [Derived] Lowe JR, Rieger RE, Moss NC, Yeo RA, Winter S, Patel S, Phillips J, Campbell R, Baker S, Gonzales S, Ohls RK. Impact of Erythropoiesis-Stimulating Agents on Behavioral Measures in Children Born Preterm. J Pediatr. 2017 May;184:75-80.e1. doi: 10.1016/j.jpeds.2017.01.020. Epub 2017 Feb 6. PMID 28185625
- [Derived] Ohls RK, Cannon DC, Phillips J, Caprihan A, Patel S, Winter S, Steffen M, Yeo RA, Campbell R, Wiedmeier S, Baker S, Gonzales S, Lowe J. Preschool Assessment of Preterm Infants Treated With Darbepoetin and Erythropoietin. Pediatrics. 2016 Mar;137(3):e20153859. doi: 10.1542/peds.2015-3859. Epub 2016 Feb 15. PMID 26908704

RESULTS

PARTICIPANT FLOW:
Groups:
- Preterm ESA Recipients: infants 500-1250 grams who received erythropoietin (400 units/kg 3x/week) or darbepoetin (10 micrograms/kg 1x/week), from the first week of life through 35 weeks corrected gestation
- Term Controls: Term infants with normal delivery
- Preterm Controls: infants 500-1250 grams who received placebo (sham doing) three times a week from the first week of life through 35 weeks corrected gestation
Period: Overall Study
Arm/Group | Preterm ESA Recipients | Term Controls | Preterm Controls
Started | 39 | 24 | 14
Completed | 39 | 21 (3 subjects in this arm were not seen at the second visit.) | 11 (3 subjects in this arm were not seen at the second visit)
Not Completed | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Preterm ESA Recipients: children 3.5-4 years of age who received ESAs during hospitalization
- Preterm Controls: children 3.5-4 years of age who received placebo during hospitalization
- Term Controls: healthy children 3.5-4 years of age born term
- Total: Total of all reporting groups
Arm/Group | Preterm ESA Recipients | Preterm Controls | Term Controls | Total
Number analyzed (Participants) | 39 | 14 | 24 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 14 | 24 | 77
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 47 [44 to 50] | 48.5 [45.5 to 51.5] | 45.5 [41.5 to 49.5] | 47 [43 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 14 | 37
  Male | 22 | 8 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 14 | 34
  Not Hispanic or Latino | 24 | 9 | 10 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 3 | 3 | 14
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 26 | 11 | 20 | 57
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 14 | 24 | 77

OUTCOME MEASURES:

1. Primary Outcome: Full Scale IQ, Performance IQ, Verbal IQ, Executive Function
Description: Infants who received ESAs during their initial hospitalization will perform significantly better on measures of the Wechsler Preschool and Primary Scale of Intelligence (WPPSI) full scale IQ, performance IQ, verbal IQ, and executive function. Scores are standardized, 100 is an average score with a standard deviation of 15. Higher scores are better. Test scores range from 41 to 160.
Time Frame: 42-48 months and 66-72 months
Population: Subjects were seen around 4 years and 6 years of age. Initial numbers of subjects seen at 4 years were: Placebo group (14), ESA (39), Term (24). Numbers of subjects ween at 6 years were: Placebo (11), ESA (39), Term (21).
Measure: Mean (Standard Deviation); unit: standardized score on a scale
Groups:
- Placebo Group: 3.5-4 year olds who received placebo during hospitalization
- ESA Recipients: subjects received ESAs during their initial hospitalization
- Term Controls: children who were born healthy at term
Arm/Group | Placebo Group | ESA Recipients | Term Controls
Number analyzed (Participants) | 14 | 39 | 24
standardized score on a scale
  full scale IQ at 4 years | 79 (18) | 91 (17) | 103 (13)
  verbal IQ at 4 years | 83 (17) | 92 (18) | 101 (15)
  performance IQ at 4 years | 79 (19) | 93 (17) | 104 (11)
  executive function | 91 (13) | 100 (12) | 105 (8)
  full scale IQ at 6 years: number analyzed (Participants) | 11 | 39 | 21
  full scale IQ at 6 years | 82 (17) | 94 (19) | 100 (14)
  verbal IQ at 6 years: number analyzed (Participants) | 11 | 39 | 21
  verbal IQ at 6 years | 86 (17) | 93 (19) | 98 (15)
  performance IQ at 6 years: number analyzed (Participants) | 11 | 39 | 21
  performance IQ at 6 years | 82 (15) | 97 (16) | 102 (14)
  executive function at 6 years: number analyzed (Participants) | 11 | 39 | 21
  executive function at 6 years | 92 (15) | 99 (12) | 107 (11)

ADVERSE EVENTS:
Groups:
- ESA Group: children 3.5-4 years of age who received ESAs during hospitalization
- Placebo Group: children 3.5-4 years of age who received placebo during hospitalization
- Term Group: children born healthy at term
Arm/Group | ESA Group | Placebo Group | Term Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/14 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/14 | 0/24
Other Adverse Events (participants affected / at risk) | 0/39 | 0/14 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No